CLINICAL TRIAL: NCT05218837
Title: Research Plan for Development and Validation of a Logistic Regression Derived Algorithm to Estimate the Risk of Obstetric Anal Sphincter Injury in High- and Low-risk Scenarios.
Brief Title: Development and Validation of a Logistic Regression Algorithm to Predict the Risk of Obstetric Anal Sphincter Injury.
Status: Completed | Type: Observational
Sponsor: Maria Gyhagen (Other)
Responsible Party: Sponsor-Investigator, Maria Gyhagen, Principal Investigator Maria Gyhagen MD, PhD., Sodra Alvsborgs Hospital
Organization: Sodra Alvsborgs Hospital (Other)
Other Study IDs: Prediction_OASI_2022_SWE
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Sphincter (Anal); Perineal Rupture, Obstetric
Keywords: obstetric anal sphincter injury; prediction model; predictor; nulliparous women; vaginal birth after cesarean section; vaginal delivery; national birth register
MeSH Terms: interventions — Vaginal Birth after Cesarean

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First vaginal birth: The first vaginal birth in nulliparous women
  Interventions: Other: Vaginal birth
- Vaginal birth after cesarean section (VBAC): The first vaginal birth after one or more prior cesarean sections (VBAC)
  Interventions: Other: Vaginal birth
- Second vaginal delivery: The second vaginal delivery
  Interventions: Other: Vaginal birth

INTERVENTIONS:
Other: Vaginal birth — Obstetric anal sphincter injury occurs at the final stage of vaginal delivery.

SUMMARY:
An obstetric anal sphincter injury (OASI) occurs during the final stage of a vaginal delivery. This tissue laceration, even if adequately sutured, poses a substantial threat to bowel continence in women.1,2 In a recent register-based study we showed that following an OASI at the first birth, the risk of a repeat injury almost tripled and that the long-term prevalence of fecal incontinence (FI) doubled in women with 1 OASI and tripled in those with 2 consecutive OASIs, in comparison with nulliparous women not affected by childbirth.3 Most OASIs occur seemingly by chance in the absence of known risk markers, and there is still no prediction model that is of use to avoid OASI in the clinical setting.4 Therefore, these injuries are often excused as inevitable and impossible to foresee.

The aim of this study is to develop and validate prediction models for the risk of an OASI in high- and low-risk scenarios.

DETAILED DESCRIPTION:
Research plan for development and validation of a logistic regression derived algorithm to estimate the risk of obstetric anal sphincter injury

Aim The aim of this study is to develop and validate prediction models for the risk of an OASI in high- and low-risk scenarios.

Study design The study will be restricted to cover 10 years from 2009 to 2018. The primary data source will be the Swedish Medical Birth Register (MBR). In addition, data will be retrieved from the National Patient Register, which comprises data on health care episodes in inpatient (hospital) and outpatient specialist care maintained by the Swedish National Board of Health and Welfare and the Swedish Longitudinal Integrated Database for Health Insurance and Labor Market Studies maintained by Statistics Sweden.

The following inclusion criteria will be applied:

* The 1st and the 2nd vaginal delivery, with secured information on the number of births and the mode of delivery
* Singleton pregnancies
* Gestational week ≥37+0

Three separate study cohorts are planned to be analyzed:

1. The first vaginal birth in nulliparous women (high-risk)
2. The first vaginal birth after one or more prior cesarean sections (VBAC) (high-risk)
3. The second vaginal delivery (low-risk) Women from cohort 1 may contribute with their second birth to cohort 3. The main difference between the cohorts is the additional pre-natal information available in cohorts 2 and 3, compared with cohort 1.

Definition of obstetric anal sphincter injury outcome The Swedish medical registers follow the International Classification of Diseases, 10th revision (ICD-10), for OASI. For identification of the outcome OASI, the following codes will be used.

* ICD 070.2, O70.2C, O70.2D, O70.2E, O70.2F, O70.2X (third-degree tear, which involves part of or the entire anal sphincter), and/or
* ICD O70.3 (fourth-degree tear, which extends further to the rectal mucosa) and/or
* the variable "Sphincter, (SFINKTER)" is "1"
* the surgical Diagnosis Related Groups code, MBC33 (suture of a third- or a fourth-degree perineal tear).

Predictors of obstetric anal sphincter injury The selection of candidate predictor variables for OASI will be based on our previous works on OASI, a search of systematic reviews and meta-analyses in the literature, and clinically relevant and retrievable information in the registers.

Candidate predictors:

Maternal demographics Age Weight in early pregnancy Weight gain since prior pregnancy Height Body mass index Smoking habits during pregnancy Education Income Country of birth Prior obstetric information (maternal and infant) Emergency C-section Elective C-section Apgar score Large-for-gestational-age Infant birth weight Infant head circumference Obstetric anal sphincter injury Vacuum delivery Forceps delivery Labor induction Labor augmentation Episiotomy Weight gain since prior pregnancy Maternal diseases (current) Recurrent cystitis Chronic kidney diseases Diabetes type I and II, pre- pregnancy Epilepsy Asthma Inflammatory bowel disease Systemic lupus erythematosus Hypertensive diseases Pregnancy diabetes Labor Labor induction* Labor augmentation Episiotomy Vacuum delivery Forceps delivery Epidural anesthesia* Spinal anesthesia* Infant birth characteristics Birth weight* Head circumference* Gestational age* Large-for-gestational-age* Gender* Presentation at delivery Time of day of birth

Conditional pre-natal predictors, variables in Cohort 1, which only can (or could) be determined or planned pre-birth, include maternal demographics and diseases, gestational age, fetal position, male gender, induction of labor, and, in some cases, the presence of macrosomia. *At present, the infant birth weight, head circumference, and gestational age at delivery are documented post-partum. However, the ultrasonographic biometry technique for estimating fetal weight and head circumference is developing, so we will include these variables in all models.

Statistical analysis plan

The split-sample validation approach will be used with a temporal split according to the period for birth [development/training data set 2012-2018 (~70%) vs. validation/test data set 2009-2011 (~30%)]. Logistic regression statistics will be used as the main predictor modeling tool. A model will be developed from the training dataset based on the minimization of the Bayesian Information Criteria (BIC) using the "best subset selection" approach. Model performance and stability will be evaluated using a bootstrap approach with 200 samples developing models in each sample and comparing with the model from the whole training dataset and the global model.

Non-linear effects will be evaluated using natural cubic splines with 5 knots at the 5th, 27.5th, 50th, 72.5th, and 95th percentiles. Linear and splines effects will be included simultaneously in the model selection procedure, enabling a data-driven selection between linear and non-linear trends. Transformations and cut-offs of predictor variables may be tested if needed.

The model developed on the training data will then be compared with the validation data using calibration plots. Risk scoring systems will be generated from the final models to obtain individual risk scores and predicted probabilities. Women will be divided into three risk groups: low, medium, and high risk.

Three different models per cohort will be constructed (resulting in 3x2 = 6 models).

1. Predictors known pre-pregnancy (Maternal variables)
2. Predictors known post-partum (Maternal variables + Pregnancy + Neonatal + Labour)
3. Predictors known post-partum (Maternal variables + Conditional pre-natal predictors)

ELIGIBILITY:
Inclusion Criteria:

* The 1st and the 2nd vaginal delivery, with secured information on the number of births and the mode of delivery
* Singleton pregnancies
* Gestational week ≥37+0

Exclusion Criteria:

• Preterm deliveries <37 weeks

•. Multifetal pregnancies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population studied and their obstetric data were obtained from the Swedish Medical Birth Register (MBR). The MBR, which was started in 1973, is a national register that includes more than 98% of all births in Sweden. Data from all antenatal clinics and all obstetric units are sent to the MBR at the National Board of Health and Welfare (SoS). Obstetrical parameters from the delivery were obtained from the MBR. The study will be restricted to cover 10 years from 2009 to 2018. In addition, data will be retrieved from the National Patient Register, which comprises data on health care episodes in inpatient (hospital) and outpatient specialist care maintained by SoS and the Swedish Longitudinal Integrated Database for Health Insurance and Labor Market Studies maintained by Statistics Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 800000 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Obstetric anal sphincter injury in term pregnancy ≥ 37+0 and a singleton pregnancy | 2009-2018
  The Swedish medical birth register (MBR) follow the International Classification of Diseases, 10th revision (ICD-10), for OASI. For identification of the outcome OASI, the following codes will be used.
  * ICD 070.2, O70.2C, O70.2D, O70.2E, O70.2F, O70.2X (third-degree tear, which involves part of or the entire anal sphincter), and/or
  * ICD O70.3 (fourth-degree tear, which extends further to the rectal mucosa) and/or
  * the variable "Sphincter, (SFINKTER)" is "1"
  * the surgical Diagnosis Related Groups (DRG code) is MBC33 (suture of a third- or a fourth-degree perineal tear).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gyhagen, MD, PhD, Principal Investigator
Locations (1):
- Maria Gyhagen, Borås, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bols EM, Hendriks EJ, Berghmans BC, Baeten CG, Nijhuis JG, de Bie RA. A systematic review of etiological factors for postpartum fecal incontinence. Acta Obstet Gynecol Scand. 2010 Mar;89(3):302-14. doi: 10.3109/00016340903576004. PMID 20199348
- [Result] Nilsson IEK, Akervall S, Molin M, Milsom I, Gyhagen M. Symptoms of fecal incontinence two decades after no, one, or two obstetrical anal sphincter injuries. Am J Obstet Gynecol. 2021 Mar;224(3):276.e1-276.e23. doi: 10.1016/j.ajog.2020.08.051. Epub 2020 Aug 21. PMID 32835724
- [Result] Webb SS, Hemming K, Khalfaoui MY, Henriksen TB, Kindberg S, Stensgaard S, Kettle C, Ismail KM. An obstetric sphincter injury risk identification system (OSIRIS): is this a clinically useful tool? Int Urogynecol J. 2017 Mar;28(3):367-374. doi: 10.1007/s00192-016-3125-2. Epub 2016 Sep 2. PMID 27589856
- [Result] McPherson KC, Beggs AD, Sultan AH, Thakar R. Can the risk of obstetric anal sphincter injuries (OASIs) be predicted using a risk-scoring system? BMC Res Notes. 2014 Jul 24;7:471. doi: 10.1186/1756-0500-7-471. PMID 25056485